CLINICAL TRIAL: NCT07328308
Title: Delayed Surveillance Colonoscopy Following Piecemeal EMR - a Randomized Study
Brief Title: Delayed Surveillance Colonoscopy Following Piecemeal EMR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Amir Klein MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RMB-0069-25
Record Dates: First submitted 2025-12-18; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer Prevention; Polyp Colorectal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Surveillance Group (Active Comparator): Participants undergo colonoscopy at 6, 18, and 48 months after piecemeal EMR.
  Interventions: Procedure: Colonoscopy after bowel cleansing
- Relaxed Surveillance Group (Experimental): Participants undergo colonoscopy at 12 and 48 months after piecemeal EMR.
  Interventions: Procedure: Colonoscopy after bowel cleansing

INTERVENTIONS:
Procedure: Colonoscopy after bowel cleansing — The procedure is performed by experienced endoscopists using high-definition white light and narrow-band imaging to carefully inspect the colon and assess the resection site. Biopsies are taken only if abnormal tissue or recurrence is suspected.

SUMMARY:
This multicenter, prospective, randomized non inferiority trial, conducted at four Israeli hospitals, will evaluate whether a relaxed surveillance strategy after piecemeal endoscopic mucosal resection (pEMR) of large non pedunculated colorectal polyps (LNPCPs, ≥20 mm) is as safe and effective as the current standard intensive surveillance. Approximately 760 adults undergoing complete pEMR with margin ablation will be randomized 1:1 into:

Standard Surveillance: Colonoscopy at 6, 18, and 48 months

Relaxed Surveillance: Colonoscopy at 12 and 48 months

All colonoscopies will be performed using high definition white light and narrow band imaging, with biopsies obtained only if recurrence is suspected. The investigators hypothesize that a relaxed surveillance strategy will be non inferior to the current standard intensive surveillance. If non inferiority is demonstrated, the study may support guideline changes toward reduced surveillance frequency after pEMR with margin ablation, potentially decreasing patient burden and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Undergoing pEMR of LNPCPs
* Able to provide informed consent and comply with follow-up requirements

Exclusion Criteria:

* Patients with invasive cancer identified during the index procedure
* en bloc resection
* Patients unable to attend follow-up colonoscopies due to comorbid conditions
* Patients who require additional surgery for polyp removal or other complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Rate of residual/recurrent adenoma (RRA) at first and second surveillance colonoscopy. | From patient enrollment until the end of the 48 month follow up period

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-12-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT07328308/Prot_000.pdf